CLINICAL TRIAL: NCT02765776
Title: An Observational Retrospective Database Analysis to Evaluate Raltegravir Based-regimens, Including NUC-sparing Regimens, in Aged HIV Patients (RalAge)
Brief Title: An Observational Retrospective Database Analysis to Evaluate Raltegravir Based-regimens in Aged HIV Patients (RalAge)
Acronym: RalAge
Status: Completed | Type: Observational
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Dott.ssa Gabriella D'Ettorre, MD, PhD, Azienda Policlinico Umberto I
Other Study IDs: RalAge d'Ettorre 2016
Record Dates: First submitted 2016-05-02; First posted 2016-05-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2016-05

CONDITIONS: HIV
Keywords: Anti-HIV Drugs; Raltegravir Potassium; Aged; Retrospective Study; Medical Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational retrospective cohort to describe RAL data — This is an observational retrospective cohort in real world to describe RAL data, including NUC-sparing regimens, in aged HIV patients.
  In this retrospective analysis all naïve patients on raltegravir-based regimens and all patients switched to raltegravir-based regimens will be considered. For raltegravir-based regimens the investigators mean raltegravir as third agent in a triple regimen with NRTIs and also raltegravir-based regimens in NUC-sparing therapies. Data will be collected from medical records. The Time horizon for patient follow-up for outcome is at least 12 months.

SUMMARY:
RAL is considered one of the better-tolerated antiretroviral medications, due to limited side effects and few long-term safety concerns. Five-year clinical trial outcomes and clinical experience have demonstrated durable virologic suppression in both treatment-naïve and treatment-experienced patients, including patients with extensive antiretroviral history and documented antiretroviral resistance. Studies have also exhibited low adverse effect rates and reliable long-term safety lending to improved tolerance. Several trials have evaluated the reduction in adverse effects in patients switched from various antiretroviral agents to RAL. Treatment-naïve studies have demonstrated a lipid-neutral effect in patients on RAL-containing regimens. When transitioning patients from a ritonavir-boosted PI regimen, statistically significant decreases in total plasma cholesterol, low-density lipoprotein, and triglycerides were demonstrated. Given its negligible interaction with the cytochrome P450 system, RAL displays minimal drug-drug interactions, making it a good option for ageing patients on multiple medications.

This is an observational retrospective cohort in real world to describe RAL data, including NUC-sparing regimens, in aged HIV patients. It is a phase IV study. 90 patients will be enrolled from the Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 4000 HIV patients are followed at this Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 50% of these patients are ≥ 50 years. From 10 to 12% are treated with a raltegravir based- regimen.

The primary endpoint will be the description of the proportion of participants with an HIV-1 viral load < 50 copies/mL.

The secondary endpoints will be:

* Change from Baseline in CD4+ T-cell counts, CD8 cell counts, CD4/ CD8 ratio
* Proportion of subjects with laboratory alterations
* Proportion of patients with adverse events (AE), serious adverse events (SAE), also according to their severity

DETAILED DESCRIPTION:
Objectives The primary endpoint will be the description of the proportion of participants with an HIV-1 viral load < 50 copies/mL.

The secondary endpoints will be:

* Change from Baseline in CD4+ T-cell counts, CD8 cell counts, CD4/ CD8 ratio
* Proportion of subjects with laboratory alterations
* Proportion of patients with adverse events (AE), serious adverse events (SAE), also according to their severity

Hypotheses Being this a retrospective study, a formal hypothesis is not formulated. Background and Rationale Antiretroviral therapy has changed the natural history of HIV infection. However, antiretroviral therapy must be maintained for life. Its potential long-term adverse effects may interact synergistically with the ageing process, resulting in a higher incidence of comorbidities. The increasing number of non-antiretroviral drugs used to treat comorbidities may also place the patient at a higher risk of clinically meaningful interactions. Nowadays, efficacy is well demonstrated by all antiretroviral drugs compared with previous times. In fact a substantial number of HIV-infected patients from areas where antiretroviral therapy is widely available have achieved sustained suppression of plasma HIV replication. In contrast, the contributions of antiretroviral therapy to the development and progression of comorbidities and to the risk of potentially severe interactions have gained increasing importance as HIV-infected patients are getting older. More than half of HIV-infected patients aged ≥ 50 years have been reported to suffer from two or more concomitant comorbidities. In some of these patients, maintenance of antiretroviral therapy with combinations including NRTIs or PIs may be challenging. Data on ageing HIV patients under antiretroviral therapy are lacking.

RAL is considered one of the better-tolerated antiretroviral medications, due to limited side effects and few long-term safety concerns. Five-year clinical trial outcomes and clinical experience have demonstrated durable virologic suppression in both treatment-naïve and treatment-experienced patients, including patients with extensive antiretroviral history and documented antiretroviral resistance. Studies have also exhibited low adverse effect rates and reliable long-term safety lending to improved tolerance. Several trials have evaluated the reduction in adverse effects in patients switched from various antiretroviral agents to RAL. Treatment-naïve studies have demonstrated a lipid-neutral effect in patients on RAL-containing regimens. When transitioning patients from a ritonavir-boosted PI regimen, statistically significant decreases in total plasma cholesterol, low-density lipoprotein, and triglycerides were demonstrated. Given its negligible interaction with the cytochrome P450 system, RAL displays minimal drug-drug interactions, making it a good option for ageing patients on multiple medications.

Study Design This is an observational retrospective cohort in real world to describe RAL data, including NUC-sparing regimens, in aged HIV patients. It is a phase IV study. 90 patients will be enrolled from the Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 4000 HIV patients are followed at this Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 50% of these patients are ≥ 50 years. From 10 to 12% are treated with a raltegravir based- regimen.

In this retrospective analysis all naïve patients on raltegravir-based regimens and all patients switched to raltegravir-based regimens will be considered. For raltegravir-based regimens the investigators mean raltegravir as third agent in a triple regimen with NRTIs and also raltegravir-based regimens in NUC-sparing therapies.

Raltegravir initiation is equivalent to baseline.

All consecutive patients fulfilling the following inclusion criteria are considered eligible:

* HIV-1 infected patients,
* aged ≥ 60 years old
* naive patients receiving raltegravir based-regimen, including Nuc-sparing regimens,
* experienced patients with virological suppression (HIV-1 RNA<50 copies) who had switched from any antiretroviral drug to raltegravir-based regimens (including Nuc-sparing regimens) because of toxicity, convenience or other reasons.

Data are collected from medical records. The Time horizon for patient follow-up for outcome is at least 12 months.

The following information will be extracted from the database of the Department:

* demographics (age, sex, race)
* smoking
* risk factors for HIV infection
* time from HIV-1 diagnosis (years)
* history of AIDS diagnosis
* hepatitis C virus (HCV) co-infection
* hepatitis B virus (HBV) co-infection
* presence of co-morbidities (including diabetes, hypertension, CVD, CKD, cancer, etc)
* reasons for switching to raltegravir
* time with HIV-1 RNA < 50 copies/mL before switch
* BMI
* Hematology (Hb, PLT)
* Creatinine
* eGFR (CKD-EPI formula)
* Phosphorus
* Calcium
* AST
* ALT
* alkaline phosphatase
* total, direct, indirect bilirubin
* proteinuria
* total, HDL-, LDL-cholesterol
* triglycerides
* glycemia
* HIV-RNA
* CD4+, CD8, CD4/CD8 ratio since the start of raltegravir
* previous ART regimen and number of previous antiretroviral agents.

Follow-up will count from the date of start of raltegravir to VF/TF or last available visit, whichever first occurred

AEs were classified as mild/moderate, severe or life threatening, according to DAIDS Classification. AEs were considered unrelated to RAL, possibly related or related, according to physician criteria.

Safety data will be descriptive; no comparison data will be analyzed.

Study Procedures At study visits, clinical data are collected and laboratory analyses comprising CD4+ T cell count, plasma HIV-1 RNA, blood cells, and plasma chemistry profiles, including fasting lipids (total cholesterol, high-density lipoprotein cholesterol [HDL], low- density lipoprotein [LDL] cholesterol, triglycerides) are recorded. Plasma HIV-1 RNA and all other laboratory determinations are performed locally at each site throughout the follow-up period.

Study Duration The Time horizon for patient follow-up for outcome is at least 12 months.

Statistical Analysis and Sample Size Justification Descriptive analyses

Baseline characteristics of enrolled patients will be presented as mean values ± standard deviation (SD) and median value with interquartile range, absolute frequency (relative frequency) according to the variable type and distribution.

Primary analysis The proportion of patients with an HIV-1 viral load < 50 copies/mL will be expressed as frequency and percentage. The 95% confidence intervals (CIs) of proportion and corresponding incidence rate will be calculated.

Secondary analyses The change from baseline of continuous variables will be assessed by the Student's t-test for paired data for normally distributed variables (based on the Shapiro-Wilk statistics) and the Wilcoxon signed-rank test for non normally distributes ones. All tests will be two-sided and a p-value of less than 0.05 will be considered as statistically significant.

Safety data analysis will be descriptive only. Safety data (AEs, SAEs) and laboratory alterations will be tabulated, according to their severity, for a descriptive purpose only.

Power/Sample Size:

A sample size of 90 subjects produces two-sided 95% CI with the following width: when the sample proportion of patients with an HIV-1 viral load < 50 copies/mL is between 40% and 60%, the 95% CI width is 0.2, that correspond to the possible maximum width in this study. Corresponding widths are 0.17 for a sample proportion of 0.30 (or 0.70), 0.15 for a sample proportion of 0.20 (or 0.80) and 0.13 for a sample proportion of 0.10 (or 0.90) (PASS 11. NCSS, LLC. Kaysville, Utah, USA).

Specific Drug Supply Requirements No drug supply is required

Adverse Experience Reporting Safety data will be descriptive; no comparison data will be analyzed. If adverse events will be identified they will be reported to the Italian agency for Drugs (AIFA) according to the law.

Safety Assessments For the International Conference on Harmonization (ICH), an AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.

SAE is any untoward medical occurrence or effect that at any dose:

1. Results in death;
2. Is life-threatening;
3. Requires hospitalization or prolongation of existing inpatients' hospitalization;
4. Results in persistent or significant disability or incapacity; and/or
5. Is a congenital anomaly or birth defect;
6. Is a cancer;
7. Is associated with an overdose;
8. Is an Other Important Medical Event.

Life-threatening in the definition of a serious adverse event refers to an event in which the subject was at risk of death at the time of event; it does not refer to an event which hypothetically might have caused death if it were more severe.

Medical judgment should be exercised in deciding whether an adverse event/reaction is serious in other situations. Important adverse events/ reactions that are not immediately life-threatening or do not result in death or hospitalization, but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above, should also be considered serious.

The severity of AEs will be graded according to the following definitions:

Mild: awareness of sign, symptom, or event, but easily tolerated; Moderate: discomfort enough to cause interference with usual activity and may warrant intervention; Severe: incapacitating with inability to do normal daily living activities or significantly affects clinical status, and warrants intervention Further details will be included in the study agreement.

Publication Plan

The publication plan will consider one manuscript.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients,
* aged ≥ 60 years old
* naive patients receiving raltegravir based-regimen, including Nuc-sparing regimens,
* experienced patients with virological suppression (HIV-1 RNA<50 copies) who had switched from any antiretroviral drug to raltegravir-based regimens (including Nuc-sparing regimens) because of toxicity, convenience or other reasons.

Exclusion Criteria:

* There are no exclusion criteria as retrospective study on medical records

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective analysis all naïve patients on raltegravir-based regimens and all patients switched to raltegravir-based regimens will be considered. For raltegravir-based regimens the investigators mean raltegravir as third agent in a triple regimen with NRTIs and also raltegravir-based regimens in NUC-sparing therapies.
  Raltegravir initiation is equivalent to baseline. All consecutive patients fulfilling the inclusion criteria are considered eligible.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an HIV-1 viral load < 50 copies/mL | 12 months

SECONDARY OUTCOMES:
Change from Baseline in CD4+ T-cell counts | 12 months
Change from Baseline in CD8+ t-cell counts, CD8 cell counts | 12 months
Change from Baseline in CD4/ CD8 ratio | 12 months
Proportion of patients with adverse events (AE), serious adverse events (SAE), also according to their severity | 12 months
demographics (age, sex, race) | 12 months
smoking | 12 months
risk factors for HIV infection | 12 months
time from HIV-1 diagnosis | 12 months
history of AIDS diagnosis | 12 months
hepatitis C virus (HCV) and hepatitis B virus co-infection | 12 months
presence of co-morbidities | 12 months
  including diabetes, hypertension, CVD, CKD, cancer, etc
previous ART regimen | 12 months
Number of previous antiretroviral agents | 12 months
reasons for switching to raltegravir | 12 months
time with HIV-1 RNA < 50 copies/mL before switch | 12 months
weight in kilograms | 12 months
height in meters | 12 months
BMI in kg/m^2 | 12 months
Hematology (Hb, PLT) | 12 months
Creatinine | 12 months
eGFR (CKD-EPI formula) | 12 months
Phosphorus | 12 months
Calcium | 12 months
AST and ALT | 12 months
alkaline phosphatase | 12 months
total, direct, indirect bilirubin | 12 months
proteinuria | 12 months
total, HDL-, LDL-cholesterol | 12 months
triglycerides | 12 months
glycemia in mg/dL | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella d'Ettorre, MD, PhD, Principal Investigator — Azienda Policlinico Umberto I (Rome)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Monteiro P, Perez I, Laguno M, Martinez-Rebollar M, Gonzalez-Cordon A, Lonca M, Mallolas J, Blanco JL, Gatell JM, Martinez E. Dual therapy with etravirine plus raltegravir for virologically suppressed HIV-infected patients: a pilot study. J Antimicrob Chemother. 2014 Mar;69(3):742-8. doi: 10.1093/jac/dkt406. Epub 2013 Oct 14. PMID 24128667
- [Background] Liedtke MD, Tomlin CR, Lockhart SM, Miller MM, Rathbun RC. Long-term efficacy and safety of raltegravir in the management of HIV infection. Infect Drug Resist. 2014 Mar 18;7:73-84. doi: 10.2147/IDR.S40168. eCollection 2014. PMID 24672249
- [Result] Pavone P, Giustini N, Fimiani C, Paoletti F, Falciano M, Salotti A, Di Sora F, Al Moghazi S, Mezzaroma I, Vullo V, d'Ettorre G. Long-Term Treatment With Raltegravir is Associated with Lower Triglycerides and Platelets Count in the Older HIV+ Population: Results from the Ral-Age Study. Curr HIV Res. 2017 Nov 23;15(5):355-360. doi: 10.2174/1570162X15666170927124558. PMID 28969567
- [Derived] Santinelli L, Ceccarelli G, Borrazzo C, Celani L, Pavone P, Innocenti GP, Spagnolello O, Fimiani C, Ceci F, Di Sora F, Mezzaroma I, Mastroianni CM, d'Ettorre G. Real word outcomes associated with use of raltegravir in older people living with HIV: results from the 60 months follow-up of the RAL-age cohort. Expert Rev Anti Infect Ther. 2020 May;18(5):485-492. doi: 10.1080/14787210.2020.1733415. Epub 2020 Feb 25. PMID 32096433